CLINICAL TRIAL: NCT03900780
Title: Preimplantion Genetic Testing for Aneuploidies (PGT-A) in Patients With Recurrent Implantation Failure: a Pilot RCT
Brief Title: Preimplantation Genetic Testing for Aneuploidies in Patients With Recurrent Implantation Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Brecht Geysenbergh, Principal Investigator, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S62302
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Recurrent Implantation Failure

STUDY DESIGN:
Intervention Model Description: Pilot RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PGT-A group (Experimental): ovarian stimulation, oocyte aspiration, embryo culture until the blastocyst stage (day 5/6), TE biopsy, vitrification of all embryos in the blastocyst stage, PGT-A by NGS and finally embryo transfer of genetically normal embryos in cumulative frozen-thawed embryo transfer cycles
  Interventions: Procedure: PGT-A
- Control group (Active Comparator): ovarian stimulation, oocyte aspiration, embryo culture until the blastocyst stage, fresh embryo transfer of the morphologically best embryo on day 5/6, vitrification of supernumerary embryos and embryo transfer in cumulative frozen-thawed embryo transfer cycles if not pregnant from the fresh cycle.
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: PGT-A — ovarian stimulation, oocyte aspiration, embryo culture until the blastocyst stage (day 5/6), TE biopsy, vitrification of all embryos in the blastocyst stage, PGT-A by NGS and finally embryo transfer of genetically normal embryos in cumulative frozen-thawed embryo transfer cycles
  Arms: PGT-A group
Procedure: Control — ovarian stimulation, oocyte aspiration, embryo culture until the blastocyst stage, fresh embryo transfer of the morphologically best embryo on day 5/6, vitrification of supernumerary embryos and embryo transfer in cumulative frozen-thawed embryo transfer cycles if not pregnant from the fresh cycle.
  Arms: Control group

SUMMARY:
Assessing whether Preimplantation Genetic Testing for Aneuploidy (PGT-A) can increase the ongoing pregnancy rate per transferred embryo and can decrease the time to pregnancy and miscarriage rate in patients with Recurrent Implantation Failure (RIF)

ELIGIBILITY:
Inclusion Criteria:

* Women with recurrent implantation failure (previous transfer of least 4 good quality embryos in at least 3 fresh or frozen cycles)
* BMI < 35
* Normal hysteroscopy

Exclusion Criteria:

* thin endometrium in previous cycles (<6mm), endometriosis ASRM score III-IV, premature ovarian failure (POF, Bologna criteria), abnormal karyotype, donor oocytes or embryos, PGT-M

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
OPR | at 20 weeks gestational age
  Ongoing pregnancy rate per embryo transfer

SECONDARY OUTCOMES:
IR | 2 weeks
  Implantation rate per transferred embryo

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No